CLINICAL TRIAL: NCT07092878
Title: Effects of Chamomile With L-theanine Beverage Among Young Women Experiencing Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Tan Chin Xuan, Assistant Professor, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 78-373
Record Dates: First submitted 2025-07-13; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Primary Dysmenorrhea
Keywords: primary dysmenorrhea; sleep; mood
MeSH Terms: interventions — Chamomile extract

STUDY DESIGN:
Intervention Model Description: Participants in the intervention group will consume a chamomile with L-theanine (CTT) beverage, which will contain 480 mg of chamomile extract and 200 mg of L-theanine. In contrast, those in the control group will consume a chamomile-flavored beverage (non-CTT), which will be flavored with commercial chamomile flavoring.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTT (Experimental): Participants in the intervention group will consume a chamomile with L-theanine (CTT) beverage, which contains 480 mg of chamomile extract and 200 mg of L-theanine.
  Interventions: Dietary Supplement: Chamomile (Matricaria recutita)
- Non-CTT (Placebo Comparator): Participants in the control group will consume a chamomile-flavored beverage (non-CTT), which is flavored with commercial chamomile flavoring.
  Interventions: Dietary Supplement: Chamomile

INTERVENTIONS:
Dietary Supplement: Chamomile (Matricaria recutita) — Participants in the intervention group will consume the chamomile with L-theanine (CTT) beverage, which contains 480 mg of chamomile extract and 200 mg of L-theanine.
  Arms: CTT
Dietary Supplement: Chamomile — A chamomile-flavored beverage
  Other Names: Chamomile flavored beverage
  Arms: Non-CTT

SUMMARY:
This study aims to evaluate the effects of a beverage containing chamomile and L-theanine on menstrual symptoms, pain intensity, mood, and sleep quality among young adult females with primary dysmenorrhea.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of a beverage containing chamomile and L-theanine on menstrual symptoms, pain intensity, mood, and sleep quality among young adult females with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* A VAS score of ≥4 cm for the past three consecutive menstrual cycles
* Regular monthly menstruation
* No history of allergies or psychological/gynecological illnesses
* Absence of secondary dysmenorrhea
* No current use of any medications
* No ongoing non-pharmacological management for dysmenorrhea.

Exclusion Criteria:

* Pregnant
* Breastfeeding

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Respondents who meet the following criteria are invited to participate in phase two of the study: a VAS score of ≥4 cm for the past three consecutive menstrual cycles, regular monthly menstruation, no history of allergies or psychological/gynecological illnesses, absence of secondary dysmenorrhea, no current use of any medications (including pain relievers), and no ongoing non-pharmacological management for dysmenorrhea.
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 months
  The pain intensity is assessed using the Visual Analogue Scale (VAS) and the Numeric Rating Scale (NRS). Participants mark the point on the scale (0 to 10) that best represents the average intensity of their menstrual pain. A higher score on the VAS and NRS indicates greater pain intensity.
Menstrual symptoms | 2 months
  The Cox Menstrual Symptom Scale (CMSS) is used to assess the severity of menstrual-related symptoms experienced by participants during their most recent menstrual cycle. Each item in the CMSS is rated on a scale from 0 (not noticeable), 1 (slightly bothersome), 2 (moderately bothersome), 3 (severely bothersome), to 4 (very severely bothersome).
Sleep quality | 2 months
  The Pittsburgh Sleep Quality Index (PSQI) is used to assess the sleep quality of participants during the past week. The total PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Mood | 2 months
  The Profile of Mood States (POMS) is used to assess six mood subscales (vigor, tension, depression, anger, fatigue, and confusion) of participants during the past week. Each item is rated on a 5-point Likert scale, ranging from 0 (not at all), 1 (a little), 2 (moderately), 3 (quite a lot), and 4 (extremely).

SECONDARY OUTCOMES:
Hemoglobin | 2 months
  Hemoglobin is measured in mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- UTAR, Kampar, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
This project is financially supported by a beverage company and may contain commercially sensitive data. If other researchers require the IPD, they must obtain approval from the beverage company through the principal investigator.